CLINICAL TRIAL: NCT07049783
Title: Examining the Circadian Timing Effects of the Hypotensive Response to Exercise
Acronym: XTIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Freda Patterson (Other)
Responsible Party: Sponsor-Investigator, Freda Patterson, Professor, University of Delaware
Organization: University of Delaware (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2324519-1
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Young Adults; Hypertension; Post-Exercise Hypotension; Circadian Rhythm
Keywords: Young adults; Hypertension; Post-exercise hypotension; Circadian rhythm
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning (Experimental): Exercise 10 hours after dim-light melatonin onset
  Interventions: Behavioral: Exercise
- Afternoon (Experimental): Exercise 15 hours after dim-light melatonin onset
  Interventions: Behavioral: Exercise
- Evening (Experimental): Exercise 20 hours after dim-light melatonin onset
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — A single standardized, in-lab, 30-minute monitored treadmill exercise session

SUMMARY:
The goal of this study is to learn how exercise timing affects blood pressure in adults with elevated or high blood pressure. Exercise can influence the body's natural 24-hour rhythms, including blood pressure patterns. A single exercise session can lower blood pressure for up to 24 hours, but it is not fully understood how the time-of-day for exercise affects this response. The main question this study aims to answer is:

• When the same participant exercises at different times of day (morning, afternoon, or evening), how does this affect the participant's blood pressure over the next 24 hours?

Participants will:

* Undergo an in-lab assessment of individual biological rhythm that will indicate the clock-time for an individual's biological night
* Complete 3 supervised treadmill exercise sessions

  * 1 in the biological morning (biological night + 10 hours)
  * 1 in the biological afternoon (biological night + 15 hours)
  * 1 in the biological evening (biological night + 20 hours)
* Complete a 24-hour blood pressure assessment before and after each exercise session

DETAILED DESCRIPTION:
This fully counterbalanced, within-subject, randomized crossover trial will examine the time-of-day dependent hypotensive effect of exercise in adults aged 18-39 years with elevated blood pressure or stage 1 hypertension. To examine this, participants will complete an assessment of dim-light melatonin onset (DLMO), the gold standard assessment of individual circadian phase, which will be used to subsequently prescribe three exercise sessions in the morning (10 hours after DLMO), afternoon (15 hours after DLMO), and evening (20 hours after DLMO) with 24-hour blood pressure assessment before and after each exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 Years old
* Resting blood pressure greater than or equal to 120/80 mmHg or less than 140/90 mmHg

Exclusion Criteria:

* Diagnosis or history of chronic or autoimmune disease (i.e., cardiovascular, metabolic, renal, endocrine, cancer)
* Diagnosis or history of sleep disorder (i.e., obstructive sleep apnea, insomnia, restless leg syndrome)
* Alcohol or drug dependence
* Elevated risk for sleep disorders
* Elevated risk for clinical depression
* Normotensive (blood pressure less than 120/80 mmHg) or stage 2+ hypertension (blood pressure greater than or equal to 140/90 mmHg)
* Body mass index less than 18.5 or greater than 35 kg/m2
* Self-reported use of sleep medications/supplements (e.g., melatonin)
* Self-reported use of medications influencing vascular physiology (e.g., antihypertensive medications, weight loss medications)
* Highly physically active (greater than or equal to 300 minutes moderate-to-vigorous physical activity per week)
* Currently pregnant or breastfeeding
* Current tobacco use (greater than or equal to 1 cigarette in the past month)
* Nighttime or rotating shift work within the last 3 months
* Contraindications to aerobic exercise

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Average daytime systolic blood pressure | 24-hours
  Change in average daytime systolic blood pressure (post-exercise - pre-exercise)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No